CLINICAL TRIAL: NCT04408625
Title: A Phase 1/2 Ascending Dose Study to Evaluate the Safety and Effects on Progranulin Levels of LY3884963 in Patients With Fronto-Temporal Dementia With Progranulin Mutations (FTD-GRN)
Brief Title: Phase 1/2 Clinical Trial of LY3884963 in Patients With Frontotemporal Dementia With Progranulin Mutations (FTD-GRN)
Acronym: PROCLAIM
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prevail Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J4B-MC-OKAA (PRV-FTD101)
Record Dates: First submitted 2020-05-21; First posted 2020-05-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Frontotemporal Dementia
Keywords: Fronto-Temporal Dementia; Frontotemporal Dementia; Progranulin Mutations; FTD-GRN; Gene Therapy; Dementia Gene Therapy; AAV9
MeSH Terms: conditions — Frontotemporal Dementia | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Initial Cohort - Low dose (Experimental)
  Interventions: Biological: LY3884963; Drug: Methylprednisolone; Drug: Optional Sirolimus; Drug: Optional Prednisone
- Initial Cohort - Medium dose (Experimental)
  Interventions: Biological: LY3884963; Drug: Methylprednisolone; Drug: Optional Sirolimus; Drug: Optional Prednisone
- Bridging Cohort - Low dose (Experimental): Participants enrolled in the Bridging Cohort will be assigned to either low or medium dose in an alternating manner
  Interventions: Biological: LY3884963; Drug: Methylprednisolone; Drug: Optional Sirolimus; Drug: Optional Prednisone
- Bridging Cohort - Medium dose (Experimental): Participants enrolled in the Bridging Cohort will be assigned to either low or medium dose in an alternating manner
  Interventions: Biological: LY3884963; Drug: Methylprednisolone; Drug: Optional Sirolimus; Drug: Optional Prednisone
- Cohort 5-Medium Dose (Experimental): Will enroll up to 10 participants with early phase of disease
  Interventions: Biological: LY3884963; Drug: Methylprednisolone; Drug: Optional Sirolimus; Drug: Optional Prednisone

INTERVENTIONS:
Biological: LY3884963 — Participants will receive a single dose of LY3884963, administered intra cisterna magna
Drug: Methylprednisolone — IV pulses every 2 weeks in the first 3 months.
Drug: Optional Sirolimus — At the investigators discretion following steroid tolerability issues, patients may receive a loading dose, followed by maintenance dose, followed by dose tapering; administered as concomitant medication
Drug: Optional Prednisone — If needed and at the investigator discretion, Oral Prednisone may be added to the immunosuppression regimen

SUMMARY:
Study J4B-MC-OKAA is a Phase 1/2, multi-center, open-label ascending dose, first-in-human study that will evaluate the safety and effect of intra-cisternal LY3884963 administration on progranulin protein (PGRN) levels in patients with frontotemporal dementia with progranulin mutations (FTD-GRN). Two escalating dose (low dose and medium dose) cohorts are planned, as well as one bridging cohort which will allocate patients to receive either low or medium dose. The duration of the study is 5 years. During the first year, patients will be evaluated for the effect of LY3884963 on safety, tolerability, immunogenicity, biomarkers, and efficacy. Patients will follow up for an additional 4 years to monitor safety and changes on selected biomarkers and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 30 to 85 years (inclusive), at the time of informed consent.
* Body weight range of ≥40 kg (88 lbs) to ≤110 kg (242 lb) and a BMI of 18 to 34 kg/m2.
* Has symptomatic frontotemporal dementia (FTD), including mild behavioral, cognitive, motor or language impairment per Investigator's assessment (behavioral-variant FTD, primary progressive aphasia-FTD, FTD with corticobasal syndrome, or a combination of syndromes are allowed for enrollment).
* Score ≥0.5 and ≤15 on CDR plus NACC FTLD sum of boxes (Cohorts 1-4 only). Note: In Cohort 5 only patients with CDR plus NACC FTLD with sum of boxes ≥0.5 and ≤9 AND global score of 0.5 or 1 will be enrolled.
* Stable use of background medications at least 8 weeks prior to LY3884963 dosing.
* Carrier of a pathogenic progranulin gene (GRN) mutation.
* Negative screening test for Mycobacterium tuberculosis (MTB) or documented negative MTB test within 1year prior to screening.
* Age- and gender-appropriate cancer screenings are up-to-date and completed.
* Patient and/or patient's legally authorized representative has the ability to understand the purpose and risks of the study, and provide written informed consent and authorization to use protected health information.
* Women of nonchildbearing potential must be either surgically sterile (hysterectomy, bilateral tubal ligation, salpingectomy, and/or bilateral oophorectomy at least 26 weeks before Screening) or postmenopausal, defined as spontaneous amenorrhea for at least 2 years, with follicle stimulating hormone level in the postmenopausal range at Screening based on the central laboratory's range.
* Men and women of childbearing potential (i.e., ovulating, premenopausal, and not surgically sterile) must use a highly effective method of contraception consistently and correctly for the duration of the study, including the long term follow up. Highly effective methods of contraception are those that, alone or in combination, result in a failure rate of less than 1% per year when used consistently and correctly (i.e., perfect use) and include the following for female patients of childbearing potential:

  * Combined (estrogen and progestogen containing) oral, intravaginal, or transdermal hormonal contraception associated with inhibition of ovulation.
  * Oral, injectable, or implantable progestogen-only hormonal contraception associated with inhibition of ovulation.
  * Intrauterine device.
  * Intrauterine hormone-releasing system.
  * Bilateral tubal ligation or bilateral tubal occlusion (performed at least 3 months prior to Screening).
  * Vasectomized partner (performed at least 3 months prior to Screening).
  * Sexual abstinence (no sexual intercourse), if in line with the patient's usual and preferred lifestyle.
* Acceptable forms of contraception for male patients include:

  * Sexual abstinence (no sexual intercourse), if in line with the patient's usual and preferred lifestyle.
  * History of vasectomy (performed at least 3 months prior to Screening, with documented absence of sperm in the ejaculate) in combination with condom.
  * Condom with spermicide used together with highly effective female contraceptive methods if the female partner(s) is of childbearing potential (see above for list of acceptable female contraceptive methods).

Note: Individuals who are in exclusively same sex relationships (as their preferred and usual lifestyle) are not required to use contraception.

* Men must agree to use a condom during any sexual intercourse (including male patients who have had a vasectomy) and abstain from sperm donation for the duration of the study, including long-term follow-up.
* Women must agree to abstain from egg donation for the duration of the study, including long-term follow-up.
* Women of childbearing potential cannot be pregnant or lactating/breastfeeding and must have a negative result for the serum pregnancy test (β-human chorionic gonadotropin) at Screening.
* Patient must agree to abstain from blood donation for the first year following gene transfer.
* Patient has a reliable study partner/informant (e.g. family member, friend) willing and able to participate in the study as a source of information on the patient's health status and cognitive and functional abilities.
* Patient is not dependent on a walker or wheelchair.
* Patient is living in the community (i.e. not in nursing home); some levels of assisted living may be permitted at the discretion of the investigator.
* Pneumococcal pneumonia and shingles vaccines are required within 10 years of Screening allowed to be performed during Screening but must be given at least 4 weeks prior to initiation of immunosuppressant regimen.

Exclusion Criteria:

* Diagnosis of a significant CNS (central nervous system) disease other than frontotemporal dementia (FTD) that may cause FTD symptoms or confound study objectives.
* Brain or cervical spine magnetic resonance image (MRI)/MRA imaging showing clinically significant abnormality considered to prevent intracisternal magna (ICM) injection.
* Hypersensitivity or contraindications to corticosteroid, and/or sirolimus use.
* Clinical evidence of peripheral symmetric sensory polyneuropathy (stable sensory mononeuropathies and radiculopathies are not exclusionary).
* Concomitant disease or condition within 6 months of screening that could interfere with, or treatment of which might interfere with, the conduct of the study or that would, in the opinion of the investigator, pose an unacceptable safety risk to the patient or interfere with the patient's ability to comply with study procedures
* Clinically significant laboratory test result abnormalities assessed at screening.
* Participation within 3 months prior to screening in another therapeutic investigational drug or device study with purported disease-modifying effects on FTD, unless it can be documented that the patient received placebo only.
* Any type of prior gene or cell therapy.
* Live vaccines in the 4 weeks prior to Screening. NOTE: Pneumococcal vaccine and/or shingles vaccine administration is allowed at least 4 weeks prior to initiation of immunosuppressant regimen.
* Use of blood thinners in the 2 weeks prior to screening, or anticipated use of blood thinners during the study. Antiplatelet therapies are acceptable if the patient is medically able to temporarily stop 48 hours to 7 days (depending on the antiplatelet medication used) prior to and at least 48 hours after ICM injection and LP. Note: the use of blood thinners as part of prophylaxis or treatment of an emergent VTE or another AE during the study does not exclude the patient, unless there is a baseline high risk of thromboembolic events, and use of blood thinners is highly anticipated in the opinion of the Investigator.
* Contraindications or intolerance to imaging methods (MRA, MRI, and/or computed tomography [CT]), including claustrophobia and intolerance to contrast agents used for MRI, MRA, or CT (including, but not limited to, gadolinium contrast agents and iohexol).
* Contraindications to general anesthesia or deep sedation.
* Positive urine test for drugs of abuse (including opiates, amphetamines, cocaine, barbiturates, and phencyclidine) without prescription at Screening and on Day 1.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events (AEs), Serious Adverse Events (SAEs), and Adverse Events Leading to discontinuation | 5 Years
Sum of adverse reactions (ARs) and suspected ARs | 5 years
Sum of serious ARs and serious suspected ARs | 5 years
Incidence of procedure or treatment-emergent AEs | 5 years
  Measured by brain and spine MRI
Change in AAV9, PGRN, and NfL immunogenicity in blood | Days 7, 14, and 21 and at Months 1, 1.5, 2, 3, 6, 9, 12, 18, and 24
  PGRN: progranulin protein. Measured by level of antibodies and ELISPOT
Change in AAV9, PGRN, and NfL immunogenicity in CSF | Months 2, 6, 12, 18, and 24
  Measured by levels of antibodies.
Change in PGRN levels in blood | Days 7, 14, and 21 and at Months 1, 1.5, 2, 3, 6, 9, 12, 18, and 24
Change in PGRN levels in CSF | Months 2, 6, 12, 18, and 24

SECONDARY OUTCOMES:
Change in CDR plus NACC FTLD | Months 3, 6, 9, and 12
  CDR: Clinical Dementia Rating staging instrument. NACC FTLD: National Alzheimer's Coordinating Center frontotemporal lobar degeneration domains
Change in NfL levels in blood | Days 7, 14, and 21 and at Months 1, 1.5, 2, 3, 6, 9, and 12
  NfL: neurofilament light chain
Change in NfL levels in CSF | Months 2, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Travis Lewis, MD, PhD, Study Director — Prevail Therapeutics
Locations (12):
- United States (4):
  - k2 Medical Research-Maitland, Maitland, Florida
  - PPD Phase 1 Clinic, 100 West Gore Street, Suite 202, Orlando, Florida
  - Lahey Hospital & Medical Center, 41 Burlington Mall Road, Burlington, Massachusetts
  - Hospital of the University of Pennsylvania, 3 West Gates Building, 3400 Spruce Street, Philadelphia, Pennsylvania
- Royal Prince Alfred Hospital, Brain & Mind Research Institute, 94 Mallet Street, Camperdown, New South Wales, Australia
- UZ Leuven, Neurologie Herestraat 49, Leuven, Belgium
- France (3):
  - AP-HM Hôpital de La Timone, Saint-Pierre, Marseille
  - Centre Mémoire de Ressources, Lille
  - Le Ber, Institut du Cerveau et de la Moelle Epinière, Paris
- Spain (2):
  - Hospital Clinic de Barcelona, Villaroel 170 Servicio de Neurología, Barcelona
  - Hospital Universitario de Donostia, Servicio De Neurologia, Consultas Externas Neurologia, San Sebastian, Guipúzcoa, Donostia / San Sebastian
- University College London,Queen Square, Dementia Research Building, London,, London, United Kingdom

REFERENCES:
- [Derived] Sevigny J, Uspenskaya O, Heckman LD, Wong LC, Hatch DA, Tewari A, Vandenberghe R, Irwin DJ, Saracino D, Le Ber I, Ahmed R, Rohrer JD, Boxer AL, Boland S, Sheehan P, Brandes A, Burstein SR, Shykind BM, Kamalakaran S, Daniels CW, David Litwack E, Mahoney E, Velaga J, McNamara I, Sondergaard P, Sajjad SA, Kobayashi YM, Abeliovich A, Hefti F. Progranulin AAV gene therapy for frontotemporal dementia: translational studies and phase 1/2 trial interim results. Nat Med. 2024 May;30(5):1406-1415. doi: 10.1038/s41591-024-02973-0. Epub 2024 May 14. PMID 38745011
- [Derived] De BP, Rosenberg JB, Selvan N, Wilson I, Yusufzai N, Greco A, Kaminsky SM, Heier LA, Ricart Arbona RJ, Miranda IC, Monette S, Nair A, Khanna R, Crystal RG, Sondhi D. Assessment of Safety and Biodistribution of AAVrh.10hCLN2 Following Intracisternal Administration in Nonhuman Primates for the Treatment of CLN2 Batten Disease. Hum Gene Ther. 2023 Sep;34(17-18):905-916. doi: 10.1089/hum.2023.067. PMID 37624739
- See also: Progranulin AAV gene therapy for frontotemporal dementia — https://www.nature.com/articles/s41591-024-02973-0